CLINICAL TRIAL: NCT04691973
Title: Evaluation of the Digital Health and Lifestyle Tool
Brief Title: Evaluation of Health and Lifestyle Tool
Status: Active, not recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: HealthDiabetes1
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Access to tool: Access to the digital tool. Participants use the tool at their own in addition to usual care and do the different themes that are available. They are recommended to use it at least every other week.
  Interventions: Behavioral: Health and lifestyle tool
- No access to tool: Participants are followed by their ordinary healthcare provider and are not exposed to the tool.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Health and lifestyle tool — Health and lifestyle tool used online
  Groups: Access to tool
Other: Usual care — Usual care at ordinary healthcare provider
  Groups: No access to tool

SUMMARY:
The overall aim of the study is to observe the natural pattern of usage and metabolic outcomes in patients with type 2 diabetes who had access to the new digital tool as a stand-alone support in addition to usual care. The tool is based on self-affirmation theory and has large emphasis on self-reflection to enable sustainable lifestyle changes. The changes in HbA1c, reflecting long-term blood glucose, will be evaluated in patients with type 2 diabetes. Patients are compared to controls on usual care not exposed to the tool.

DETAILED DESCRIPTION:
Considerable evidence suggest that lifestyle changes can prevent or delay the onset of type 2 diabetes, and self-care behaviors largely determine HbA1c. Modifiable lifestyle factors have been established as key drivers of disease onset, progression, and prognosis, motivating the use of "lifestyle as medicine". Despite this, a substantial number of patients with type 2 diabetes (T2D) have difficulties attaining adequate glycemic control.

Digital health tools are increasingly incorporated into diabetes care, and have the potential to improve both behavioral and clinical outcomes on a broad basis. However, low levels of uptake, reduced user engagement over time, and low acceptance among patients, raise concerns about their effectiveness. Knowledge on how to design interventions aimed at inducing change by promoting motivation and personal engagement, as well as a better understanding of patient interaction with digital health interventions, could help overcome these challenges and inform the development of a novel and effective health support.

The objective or this study is to evaluate a new web-based tool, developed at the University Gothenburg, Sweden, that aims to support patient autonomy and motivation to make sustainable lifestyle changes.

The investigators will test the hypothesis that individuals with type 2 diabetes in routine care who have access to the tool get improved HbA1c relative to baseline as compared with individuals with type 2 diabetes on usual care not exposed to the tool.

The study is an investigator-initiated single-center study conducted at Scania University Hospital, Sweden, and will follow participants over three years.

Participants with type 2 diabetes will be recruited by sending letters with study information to patients with type 2 diabetes in the region. If HbA1c is 52 mmol/mol or above participants are included and attend study visits at Scania University Hospital every three months during the first year and every sixth month during the following two years for blood sampling and physical examination.

During the first 3 months, only half of the participants get access to the tool immediately and the other half remain on usual care (randomized who get access or not). After 3 months, all participants get access to the tool and used it during an open-label observation period of up to three years.

Study visits: Every physical study visit lasts appr. 20 minutes and includes measurements of length and weight, blood pressure, and estimations of fat and muscle mass by bioimpedance. Fasting blood samples are taken for analysis of HbA1c and other cardiometabolic proteins. Participants will not receive any counselling or lifestyle advice at the study visits. Technical problems are referred to the study coordinator, who may also respond to requests to clarify content in a general manner without providing personal advice. Patients are followed by their ordinary physician throughout the study, i.e. the tool is provided on top of ordinary anti-diabetic treatment and healthcare contacts.

The tool: The tool is web-based and used via a computer or mobile phone. It is used at each individual's preferred pace but participants are recommended to login at least every other week. Every round the participants choose a themes (out of appr. 80 possible covering e.g. food, exercise, stress, self-reflection aspects), which takes appr. 15-30 minutes to complete. Participants then reflect on the content and how it could be implemented in daily life. When returning for next round participants are asked to reflect on any changes done since last time. There is no interaction between individual participants.

Statistics: The study has two primary endpoints. One primary endpoint is change of HbA1c between participants with and without access to the tool during the first 3-month period. Patients lost to follow-up will not be included in the analysis.

The standard deviation of change of HbA1c is 6 mmol/mol over 3 months. With 80% power at alpha=0.05, 142 participants are needed to each randomization arm to detect a significant difference between the groups, assuming that the true treatment effect of the intervention is 2 mmol/mol over 3 months.

Enrollment will continue until the required number of participants are reached, accounting for those lost to follow-up during the randomization period. The participants use the tool at their own pace but are within the tool recommended to complete a theme at least every other week to enable implementation of changes and maintain an awareness of the tool and its content.

As another primary endpoint, investigators will during the open-label observation period compare change of HbA1c at one year relative to baseline between patients using the tool as recommended (at least every other week) and matched controls on usual care (1:2 ratio between exposed and controls). The controls are matched on gender, age, BMI and HbA1c from existing clinical registries in the region.

The standard deviation of DeltaHbA1c is 7 mmol/mol over one year. With 80% power at alpha=0.05, 24 participants using the tool as recommended and 48 matched controls are needed to detect a significant difference between the groups, assuming that the true treatment effect of the intervention is 5 mmol/mol.

Subanalysis of MOD patients A data-driven cluster analysis of 9,000 diabetes patients has been performed in the ANDIS registry in Sweden based on six variables measured at diagnosis: GAD antibodies, age, BMI, HbA1c (reflecting long-term blood glucose), HOMA2-B (reflecting insulin secretion) and HOMA2-IR (reflecting insulin resistance). Four clusters of T2D patients were highlighted, each with different characteristics and risk of complications. One of these cluster, MOD (Mild Obesity-related Diabetes), is characterized by high BMI and insulin resistance but relatively well-preserved insulin secretion. It has been suggested that patients with MOD characteristics would benefit particularly from lifestyle changes. The investigators therefore hypothesize that patients with MOD characteristics would benefit particularly well from the intervention. As a subanalysis the investigators will analyse the interaction between MOD/non-MOD subgroup and exposure to the intervention using a linear model with a term for the cluster variable, a term for the exposure to the intervention and an interaction term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes at or above 35 years of age
* HbA1C at 52 mmol/mol or above
* Diagnosis of diabetes mellitus was based on prior documentation or treatment with anti-hyperglycemic medication
* written informed consent.

Exclusion Criteria:

* type 1 diabetes, MODY or secondary diabetes
* conditions or treatments that in the judgement of the Investigator could affect the study evaluation
* connection with the study team, funders, authorities, universities or other public or private bodies in such a way that specific interests in the study outcomes could be suspected.

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with type 2 diabetes, independent of disease duration or treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin at 3 months | 3 months
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at 3 months relative to baseline compared between participants with access to the tool and on usual care.
Change of long-term blood glucose concentration measured as glycated hemoglobin at one year | One year of the open-label observation period
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at one year relative to baseline between participants who use the tool as recommended and matched controls on usual care

SECONDARY OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin at three years | Up to three years of the open-label observation period
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at three years relative to baseline between participants who use the tool as recommended and matched controls on usual care
Body weight | 1 year
  Body weight between groups
Fat mass | 1 year
  Fat mass as estimated by bioimpedance
Muscle mass | 1 year
  Muscle mass as estimated by bioimpedance
Insulin resistance | 1 year
  Insulin resistance measured as Homeostatic model assessment (HOMA-IR)
Total Cholesterol concentration in plasma | 1 year
  Total Cholesterol concentration in plasma between groups
Low-density lipoprotein Cholesterol concentration in plasma | 1 year
  Low-density lipoprotein (LDL) Cholesterol concentration in plasma between groups
High-density lipoprotein Cholesterol concentration in plasma | 1 year
  High-density lipoprotein (HDL) concentration in plasma between groups
Triglyceride concentration in plasma | 1 year
  Triglyceride concentration in plasma between groups
Fasting blood glucose concentration | 1 year
  Fasting blood glucose concentration between groups
Systolic blood pressure | 1 year
  Systolic blood pressure between groups
Diastolic blood pressure | 1 year
  Diastolic blood pressure between groups
Quality of life estimated by 5-level European Quality-of-life (EQ-5D-5L) questionnaire score | 1 year
  Quality of life estimated by 5-level European Quality-of-life (EQ-5D-5L) questionnaire score between groups. Score is from 0 to 1 with 1 meaning highest quality of life
Physical activity in calories per day | 3 years
  Physical activity in calories per day estimated by International Physical activity questionnaire between users of the tool and controls on usual care. Score measures calorie consumption and ranges from 0 to unlimited
Insulin secretion | 1 year
  Insulin secretion estimated by Homeostatic model assessment (HOMA-B)

OTHER OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin in participants with and without Mild Obesity-related Diabetes, respectively. | 3 months and 1 year
  As a subanalysis we will analyse the effect of the tool specifically on patients with Mild Obesity-related Diabetes (MOD). This will be analysed by a formal interaction test between MOD and non-MOD participants with or without access to the tool by using a linear model with a term for MOD/non-MOD, a term for access/non-access to the tool and an interaction term.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Prof, Principal Investigator — Region Skåne
Locations (1):
- Clinical Research Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared after deidentification.
Time Frame: Data will be available after publication.
Access Criteria: To researchers who provide a methodologically sound proposal in order to achieve the aims of that proposal. Proposals should be directed by email to internetverktyg@gu.se

REFERENCES:
- [Derived] Dwibedi C, Mellergard E, Gyllensten AC, Nilsson K, Axelsson AS, Backman M, Sahlgren M, Friend SH, Persson S, Franzen S, Abrahamsson B, Carlsson KS, Rosengren AH. Effect of self-managed lifestyle treatment on glycemic control in patients with type 2 diabetes. NPJ Digit Med. 2022 May 11;5(1):60. doi: 10.1038/s41746-022-00606-9. PMID 35545657